CLINICAL TRIAL: NCT05470088
Title: Magnetic Resonance Imaging Neuroanatomical Study of Patients with an Autism Spectrum Disorder, Their Relatives and Typically Developing Subjects.
Brief Title: MRI Study of Subjects with ASD, Their Relatives and TD
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: APHP (Other); Institut Pasteur (Industry); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-90; 2017-A02356-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: neuroimaging; mri; phenotype; heritability; genes
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Neuroimaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subjects with Autism Spectrum Disorders
  Interventions: Other: Neuroimaging (MRI)
- Relatives of subjects with Autism Spectrum Disorders
  Interventions: Other: Neuroimaging (MRI)
- Typically developing subjects
  Interventions: Other: Neuroimaging (MRI)

INTERVENTIONS:
Other: Neuroimaging (MRI) — Multimodal magnetic resonance imaging

SUMMARY:
This project is structured around a central study called "Study of genetic factors involved in autism and related conditions ("Genes and Autism" study, sponsor: INSERM). This study explores clinical and genetic aspects of ASD (autism spectrum disorders) and is complemented with several ancillary studies (such as this one) which will use the data of the main study and will allow an extensive review of phenotypes associated with ASD.

In this ancillary study, we will go on the acquisition of anatomical, diffusion and functional MRI in subjects with ASD, relatives and controls. Our group has already performed several neuroanatomical studies of ASD. IWe recruited since 2010 more than 600 subjects (proponents, relatives and controls) to better understand the implication of brain abnormalities in ASD.

This study involves specialized teams in neuroiamging based at INSERM, NeuroSpin (CEA), Robert Debré Hospital (APHP) and Pasteur Institute

Our main objective is to identify structural, connectivity and functional peculiarities in subjects with ASD

Secondary objectives include:

* the identification of familial heritability patterns of ASD
* correlate data obtained in brain imaging with genetic data
* assess specificity and statistical reproducibility of the obtained results

ELIGIBILITY:
Inclusion Criteria:

* for patients:

  * being included in the main study "C16-89 - Study of genetic factors involved in ASD and related disorders"
  * having an ASD fulfilling DSM-5 diagnostic criteria (APA, 2012). Diagnosis will be done by a clinical expert, with the support of structured instruments (ADI-R, ADOS-2)
  * having at least 24 Months
  * being affiliated with the French health insurance
  * having signed the informed consent (by proposant or by legal tutors if the subject is <18 or under legal custody)
* for relatives

  * being included in the main study "C16-89 - Study of genetic factors involved in ASD and related disorders"
  * having at least 24 Months
  * being affiliated with the French health insurance
  * having signed the informed consent (by proposant or by legal tutors if the subject is <18 or under legal custody)
* for controls

  * being included in the main study "C16-89 - Study of genetic factors involved in ASD and related disorders"
  * having at least 24 Months
  * being affiliated with the French health insurance
  * having signed the informed consent (by proposant or by legal tutors if the subject is <18 or under legal custody)

Non-inclusion criteria:

* for all subjects

  * severe mental retardation (IQ<35 or developmental age<18 months)
  * medical condition (either psychiatric or physical) not compatible with an inclusion
  * MRI counter indication
  * Current pregnancy or breastfeeding, assessed by questionnaire
  * Not willing to be informed of a brain abnormality diagnosed with MRI
* for the relatives

  *discovery of non filiation during the genetic analyses
* for controls

  * Neurological history (except mental retardation)
  * Personal history of (checked with DIGS for Adults, Diagnostic Interview for Genetic Studies, Numberger et coll., 1994, or Kiddie SADS, Kiddie Schedule for Disorders and Schizophrenia for School Age Children, Orvaschel et coll., 1982): schizophrenia, addiction, bipolar disorder, recurrent depression (> 2 episodes lifetime), severe, not stabilized anxiety disorder, history of episodes of epilepsy, significant inflammatory disease of immunosuppressive medication

Exclusion Criteria:

* for patients: ASD diagnosis not confirmed by assessments after the inclusion
* for all subjects: discovery of a counter indication to MRI during the exam (e.g. claustrophobia)

Min Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of subjects above 24 months (no upper limit of age):
  * subjects with ASD
  * relatives of subjects with ASD
  * typically developing controls
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-13 (Actual); Primary Completion 2037-03-13 (Estimated); Study Completion 2039-09-13 (Estimated)

PRIMARY OUTCOMES:
3DT1 MRI derived variables | Day 0
  Cortical folding Cortical thickness Cortical surface Cortical, white matter and subcortical volumes
Resting state fMRI derived variables | Day 0
  Whole-brain BOLD signal correlations
Task based fMRI derived variables | Day 0
  BOLD activation signals BOLD signal correlations
Diffusion MRI derived variables | Day 0
  Fractional anisotropy and mean diffusivity NODDI derived variables
quantitative T1 and quantitative T2 MRI | Day 0
  Myelin Water Fraction

CONTACTS AND LOCATIONS:
Overall Officials: Richard Delorme, M.D, Ph.D, Principal Investigator — APHP, France; Josselin Houenou, M.D, Ph.D, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - NeuroSpin neuroimaging platforme, Gif-sur-Yvette
  - APHP, Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: Undecided